CLINICAL TRIAL: NCT01898416
Title: A PHASE 2, SINGLE CENTRE, SINGLE ARM STUDY TO DETERMINE THE EFFICACY AND SAFETY OF 5- ALA POHOTODYNAMIC THERAPY AS ADJUVANT THERAPY AFTER SURGICAL DISSECTION IN PATIENTS WITH DESMOID TUMORS.
Brief Title: Safety and Efficacy Study Using 5-ALA Oral Administration as an Adjuvant Therapy on the Rate of Local Tumor Recurrence in Patients Who Have Desmoids Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: michal roll (Other Government)
Responsible Party: Sponsor-Investigator, michal roll, Director research and development department, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-11-JB-558-CTIL
Record Dates: First submitted 2013-06-26; First posted 2013-07-12 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: The Aim of the Study is to Evaluate the Efficacy of Photodynamic Therapy as an; Adjuvant Therapy on the Clinical Outcome of Patients With Desmoid Tumors After; Surgical Resection
MeSH Terms: interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5-AminoLevulinicc Acid (Experimental): consists of 60mg/kg 5-ALA prepared solution given orally, 3-5 hours before induction of anesthesia and surgical tumor resection. Red light laser given by a Dye laser system, wave length of 635nm, in s dose of 150J/cm for 2000 seconds (33 minutes) will be given to tumor bed. In the case of positive margins (for tumor presence), a second surgical intervention followed by second 60mg/kg 5-ALA administration will be performed.
  Interventions: Drug: 5-AMINOLEVULINIC ACID (5-ALA), is a non fluorescent prodrug.

INTERVENTIONS:
Drug: 5-AMINOLEVULINIC ACID (5-ALA), is a non fluorescent prodrug. — 60 mg/kg 5-ALA prepared solution given orally, 3-5 hours before induction of anesthesia.
  Red light laser given by a Dye laser system, wave length of 635nm, in s dose of 150J/cm for 2000 seconds (33 minutes) will be given to tumor bed. In case of positive margins a second operation and 5-ALA administration or irradiation will be given.

SUMMARY:
The purpose of this study is to evaluate the efficacy of preoperative 5-ALA oral administration and subsequently intraoperative tumor bed phototherapy with red light laser, as an adjuvant therapy on the 3 years rate of local tumor recurrence in patients with desmoid tumors. To evaluate the Safety of 5-ALA administration. 5 years local recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a resectable histologically confirmed desmoid tumor.
2. Previously treated (by chemotherapy, irradiation or surgery) patients are eligible.
3. Age > 18 years
4. Signed informed consent prior to patient recruitment. -

Exclusion Criteria:

1. Hepatic enzymes or bilirubin > 2X upper limit of normal.
2. Serum creatinine > 2.5 x upper limit of normal.
3. Suspected /documented metastatic disease.
4. Active or uncontrolled infections.
5. Active second malignant disease (excluding non-melanoma skin cancer, or in situ cervix or breast carcinoma) < 2 years prior to the study.
6. Use of other investigational agents < 30 days prior to the study.
7. Patients who are mentally or physically unable to comply with all aspects of the study.
8. Any serious medical condition, including the presence of laboratory abnormalities, which places the subject at an unacceptable risk if he or she participates in this study or confounds the experimental ability to interpret data from the study.
9. Pregnant or lactating females.
10. Known intolerance or allergy to 5-ALA
11. Suspicious or documented acute or chronic porphyria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-06; Primary Completion 2023-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is a binary variable where each patient is classified as a recurrence or a not recurrence case and will be determined by calculating the proportion of recurrence versus non recurrence rates | three years

SECONDARY OUTCOMES:
To assess the safety of study drug administration in the study population. To assess the 5 years local recurrence rate. | five years
  Data from all subjects who receive any study drug will be included in the safety analyses. The severity of the toxicities will be graded according to the NCI CTCAE whenever possible. Adverse events will be summarized by worst NCI CTC grade. Adverse events classified as NCI CTCAE Grade 3 or Grade 4, study-drug-related events, and serious adverse events will be summarized separately. Laboratory data will be graded according to NCI CTCAE severity grade.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Bickels, MD/PhD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (2):
- Israel (2):
  - Tel Aviv sourasky medical center, Tel Aviv, Israel
  - The Aviv Sourasky Medical Center, Tel Aviv, Israel